CLINICAL TRIAL: NCT02604134
Title: Medical Management of Caries in the Primary Dentition Using Silver Nitrate: A Pilot Study
Brief Title: Medical Management of Caries in the Primary Dentition Using Silver Nitrate
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arwa Owais (Other)
Collaborators: Delta Dental of Iowa (Other)
Responsible Party: Sponsor-Investigator, Arwa Owais, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201406792
Record Dates: First submitted 2015-10-28; First posted 2015-11-13 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Dental Caries
Keywords: silver nitrate; children; dental caries; medical management; quality of life
MeSH Terms: conditions — Dental Caries | interventions — Fluorides; Silver Nitrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the radiographic progression of caries is assessed by a masked investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional treatment group (Other): The child will receive a prophylaxis and fluoride varnish. Parents will fill out a parent and a child questionnaire.
  Interventions: Procedure: Prophylaxis; Drug: Fluoride varnish
- Silver Nitrate group (Other): The child will receive a prophylaxis, then silver nitrate and then fluoride varnish. Parents will fill out a parent and a child questionnaire.
  Interventions: Procedure: Prophylaxis; Drug: Fluoride varnish; Drug: Silver Nitrate

INTERVENTIONS:
Procedure: Prophylaxis — A dental prophylaxis is a cleaning procedure performed to thoroughly clean the teeth. Prophylaxis is an important dental treatment for halting the progression of periodontal disease and gingivitis.
  Other Names: Prophy
Drug: Fluoride varnish — Fluoride varnish is a highly concentrated form of fluoride which is applied to the tooth's surface, by a dentist, dental hygienist or other health care professional, as a type of topical fluoride therapy.
  Other Names: Fluoride
Drug: Silver Nitrate — a small amount will be applied to the tooth via a cotton applicator. Silver nitrate is a colorless, odorless, transparent solution used as an escharotic, dehydrating and sclerosing agent.
  Arms: Silver Nitrate group

SUMMARY:
This pilot trial compares conventional restorations with a new strategy based on the medical management of caries using silver nitrate and fluoride varnish with no restorations.

DETAILED DESCRIPTION:
This is a two-arm, parallel group, patient-randomized controlled pilot trial. Children with at least one primary tooth where caries extends into dentine. Children will be randomized and treated according to one of two treatment approaches;(1) conventional caries management with best practice prevention, or (2) medical management of caries using silver nitrate with best practice prevention.

Baseline measures and outcome data (at treatment/review during two year follow-up) are assessed through direct reporting, clinical examination including blinded radiographic assessment, and child/parent questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Presense of one or more cavitated carious lesions in the primary dentition, extending into dentin but not encroaching on the pulp.
* Absense of any spontaneous or elicited pain due to caries, or signs of pulpal infection in response to any of the carious lesions in the primary dentition to be included in the study

Exclusion Criteria:

* Hereditary developmental defects of the teeth such as Amelogenesis Imperfecta and Dentinogenesis Imperfecta
* Medical conditions that prevent treatment of the child in the outpatient clinic. These conditions include severe bleeding disorders, cardiac problems and mental disabilities that prevent child from communication with the research team.
* Known allergy/sensitivity to any of the dental materials.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2014-07; Primary Completion 2017-08-24 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Change in baseline Caries Experience and activity (Incidence of caries in primary teeth) | through study completion, for 2 years
  Detailed measurements of caries experience will be recorded at baseline and annual caries examination using EC4

SECONDARY OUTCOMES:
Caries activity in primary teeth | through study completion, for 2 years
  Detailed measurements of caries activity will be recorded at baseline and annual caries examination using Nyvad scores.

OTHER OUTCOMES:
Pain (toothache) and/or infection in primary teeth | through study completion, for 2 years
  Assessments for pain from toothache will be made at each visit throughout the patient's participation in the trial using the Dental Discomfort Questionnaire completed by the parents.
Patient quality of life | through study completion, for 2 years
  Quality of life will be assessed through direct reporting by parents and children about pain and related activities
Cost-effectiveness | through study completion, for 2 years
  Cost-effectiveness for both groups will be calculated and compared
Acceptability of treatment strategies by parents and children | through study completion, for 2 years
  Acceptability is checked throughout the whole period of the study every time the patient comes in for a recall

CONTACTS AND LOCATIONS:
Overall Officials: Arwa I Owais, BDS, MS, Principal Investigator — Associate Profesor in Pediatric Dentistry; MIchael Kanellis, DDS, MS, Principal Investigator — Professor in Pediatric Dentistry & Dean for Patient Cares
Locations (1):
- UIowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duffin S. Back to the future: the medical management of caries introduction. J Calif Dent Assoc. 2012 Nov;40(11):852-8. PMID 23270129
- [Background] Klein U, Kanellis MJ, Drake D. Effects of four anticaries agents on lesion depth progression in an in vitro caries model. Pediatr Dent. 1999 May-Jun;21(3):176-80. PMID 10355008
- [Background] Peng JJ, Botelho MG, Matinlinna JP. Silver compounds used in dentistry for caries management: a review. J Dent. 2012 Jul;40(7):531-41. doi: 10.1016/j.jdent.2012.03.009. Epub 2012 Apr 3. PMID 22484380
- [Background] Schwendicke F, Stolpe M, Innes N. Conventional treatment, Hall Technique or immediate pulpotomy for carious primary molars: a cost-effectiveness analysis. Int Endod J. 2016 Sep;49(9):817-826. doi: 10.1111/iej.12537. Epub 2015 Sep 19. PMID 26331379
- [Background] Innes NP, Stewart M. The Hall Technique, a Simplified Method for Placing Stainless Steel Crowns on Primary Molars, may be as Successful as Traditionally Placed Crowns. J Evid Based Dent Pract. 2015 Jun;15(2):70-2. doi: 10.1016/j.jebdp.2015.03.008. Epub 2015 Mar 28. No abstract available. PMID 25987388
- [Background] Keightley A, Clarkson J, Maguire A, Speed C, Innes N. Participant recruitment to FiCTION, a primary dental care trial - survey of facilitators and barriers. Br Dent J. 2014 Nov;217(10):E22. doi: 10.1038/sj.bdj.2014.1009. PMID 25415040
- [Background] Santamaria R, Innes N. Trial shows partial caries removal is an effective technique in primary molars. Evid Based Dent. 2014 Sep;15(3):81-2. doi: 10.1038/sj.ebd.6401044. PMID 25343394
- [Background] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Splieth CH. Caries management strategies for primary molars: 1-yr randomized control trial results. J Dent Res. 2014 Nov;93(11):1062-9. doi: 10.1177/0022034514550717. Epub 2014 Sep 12. PMID 25216660
- [Result] Lamont T, Schwendicke F, Innes N. Why we need a core outcome set for trials of interventions for prevention and management of caries. Evid Based Dent. 2015 Sep;16(3):66-8. doi: 10.1038/sj.ebd.6401109. No abstract available. PMID 26492796
- [Result] Schwendicke F, Lamont T, Innes N. Outcomes in Trials for Management of Caries Lesions (OuTMaC): protocol. Trials. 2015 Sep 7;16:397. doi: 10.1186/s13063-015-0927-3. PMID 26346538